CLINICAL TRIAL: NCT02671149
Title: How do Small Changes in Hydration Influence Cognition: A Mechanistic Investigation
Brief Title: The Effect of Small Changes in Hydration on Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Responsible Party: Principal Investigator, Dr Hayley Young, Dr, Swansea University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HYD01
Record Dates: First submitted 2015-09-22; First posted 2016-02-02 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Cognition; Hydration
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drink water (Experimental): Participants will receive two 150ml drinks of water during the dehydration protocol
  Interventions: Dietary Supplement: Water
- Drink nothing (No Intervention): Participants will drink nothing during the dehydration protocol

INTERVENTIONS:
Dietary Supplement: Water — Participants will receive two cups of 150ml plain water
  Arms: Drink water

SUMMARY:
The aim of this study is to determine whether drinking plain water when mildly dehydrated benefits cognitive performance and mood. Volunteers undergo a dehydration protocol designed to result in minor dehydration. While some participants receive two 150ml drinks of water others do not. Differences in cognitive functioning are assessed.

DETAILED DESCRIPTION:
As an essential nutrient, an inadequate intake of water has negative consequences: without a source of water death will occur in days. When Benton and Young (2015) reviewed the topic they concluded that in healthy adults, mild dehydration (in the range of a loss of 2% body mass) had been found to adversely influence mood and cognition. However, it is unclear at what degree of hypohydration these effects begin to emerge.

This study was designed to determine whether small changes in hydration, of the level that might occur on a day to day basis, influence cognition and mood. During a dehydration protocol (sitting in a room heated to 30 degrees for four hours) young adult participants receive either drink two 150ml cups of water or nothing. Effects on memory, attention and mood are monitored.

ELIGIBILITY:
Inclusion Criteria:

* In good general health i.e. no major health condition such as diabetes
* BMI < 30

Exclusion Criteria:

* Not on blood pressure medication or blood thinning medication such as aspirin - No learning difficulty such as dyslexia
* Diabetes
* Gastro-intestinal disease
* High BMI
* Cholesterol and BP
* Smoker
* Dyslexic/dyspraxic
* Depression or history of depression or other psychiatric disorder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Episodic memory - list of 30 words | change from 0 to 180 minutes after the start of the dehydration protocol
  Participants listen to a list of 30 words presented using a tape recorder. The words are of similar difficulty and matched for the number of syllables and frequency with which they occur in English. The subjects are asked to recall and write down as many words as possible. The difference in the total number of words remembered from baseline (before the intervention) is analysed.
Focused attention - Eriksen Flanker Task | change from 0 to 180 minutes after the start of the dehydration protocol
  The Arrow Flankers test measures the ability to direct attention and ignore peripheral information. Participants are required to indicate whether the middle arrow is pointing to the right or left by pressing the corresponding arrow on the keyboard. Either side of the central arrow are distractors. Both the average reaction times (in milliseconds) and accuracy are recorded. The difference in performance from baseline (before the intervention) is analysed.

SECONDARY OUTCOMES:
Thirst (Participants rate their thirst) | change from 0 to 180 minutes after the start of the dehydration protocol
  Participants rate their thirst

OTHER OUTCOMES:
Amount of weight lost due to dehydration protocol | 180 minutes
  participants will be weighed at the start and end of the dehydration protocol and % weight loss calculated
Body temperature | 180 minutes
  Change in body temperature will be monitored throughout
Urine Osmolality | 180 minutes
  Urine samples will be collected at the start and end of the procedure so that changes in osmolality can be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Swansea University, Swansea, West Glamorgan, United Kingdom

REFERENCES:
- [Background] Benton D, Young HA. Do small differences in hydration status affect mood and mental performance? Nutr Rev. 2015 Sep;73 Suppl 2:83-96. doi: 10.1093/nutrit/nuv045. PMID 26290294
- [Derived] Benton D, Jenkins KT, Watkins HT, Young HA. Minor degree of hypohydration adversely influences cognition: a mediator analysis. Am J Clin Nutr. 2016 Sep;104(3):603-12. doi: 10.3945/ajcn.116.132605. Epub 2016 Aug 10. PMID 27510536